CLINICAL TRIAL: NCT02714517
Title: Efficacy of Hydrotherapy in Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: idrokinesi.neuropatie
Record Dates: First submitted 2016-03-10; First posted 2016-03-21 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Hydrotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- hydrotherapy (Experimental): patients receive daily conventional physiotherapy and three 30- minutes sessions of in- water exercises per week, for four weeks
  Interventions: Other: hydrotherapy
- controls (Active Comparator): patients receive daily conventional physiotherapy and three 30- minutes sessions of on- land exercises per week, for four weeks
  Interventions: Other: on land therapy

INTERVENTIONS:
Other: hydrotherapy — 30 minutes sessions of physiotherapy exercises in heated pool (32°C), three times per week for four weeks
  Arms: hydrotherapy
Other: on land therapy — 30 minutes sessions of physiotherapy exercises on land, three times per week for four weeks
  Arms: controls

SUMMARY:
The purpose of the study is to evaluate the efficacy of hydrotherapy on pain and balance in patients affected by neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by peripherical neuropathy able to walk

Exclusion Criteria:

* pain of water
* medical contraindications at treatment in heated swimming pool

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
balance change assessed using Berg Balance Scale | 0 and 4 weeks
disability change assessed using Functional Independence Measure scale | 0 and 4 weeks
gait change assessed using Dynamic Gait Index scale | 0 and 4 weeks
gait change assessed using Functional Ambulation Classification scale | 0 and 4 weeks
pain change assessed using Overall Neuropathy Limitation Scale | 0 and 4 weeks
disability change assessed using Neuropathy Pain Scale | 0 and 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale generale di zona Moriggia Pelascini, Gravedona Ed Uniti, CO, Italy